CLINICAL TRIAL: NCT06353373
Title: Smart Technology Facilitated In-hospital Venous Thromboembolism Prophylaxis Based on Bundled Evidence-based Prevention Strategies: the SmaVTE-BEST Study
Brief Title: Smart Technology Facilitated Venous Thromboembolism Prophylaxis Based on Bundled Evidence-based Prevention Strategies
Acronym: SmaVTE-BEST
Status: Not yet recruiting | Type: Observational
Sponsor: Navy General Hospital, Beijing (Other)
Responsible Party: Sponsor
Other Study IDs: HZKY-PJ-2024-7
Record Dates: First submitted 2024-04-01; First posted 2024-04-09 (Actual); Last update posted 2024-04-09 (Actual); Status verified 2024-03

CONDITIONS: Venous Thromboembolism; Clinical Decision Support Systems; Digital Health
Keywords: Venous Thromboembolism; Clinical Decision Support Systems; Prophylaxis
MeSH Terms: conditions — Venous Thromboembolism

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Pre-Modified DeVTEcare Group: In our hospital, routine use of DeVTEcare system (a CDSS for VTE risk assessment and integrated care) for in-hospital management of VTE has been launched since 2021. By retrospectively collecting information on discharged patients, all patients discharged from our hospital between April 2023 and April 2024 will be included in the pre-modified DeVTEcare group.
- Post-Modified DeVTEcare Group: The modified DeVTEcare system, which incorporates bundled guideline-based VTE prevention measures, will be utilized to assist healthcare providers in VTE prophylaxis after September 2024. By retrospectively collecting information on discharged patients, all patients discharged from our hospital between September 2024 and February 2025 will be included in the post-modified DeVTEcare group.
  Interventions: Other: Application of the modified DeVTEcare system

INTERVENTIONS:
Other: Application of the modified DeVTEcare system — The modified DeVTEcare system, which incorporates bundled guideline-based VTE prevention measures, will be utilized to assist healthcare providers in VTE prophylaxis after September 2024.
  Groups: Post-Modified DeVTEcare Group

SUMMARY:
Venous thromboembolism (VTE) is the third leading cause of cardiovascular disease deaths globally, and its incidence is increasing over the years. Hospital-acquired VTE accounts for approximately 75% of all deaths attributed to VTE. However, only half of patients with indications for VTE prophylaxis take preventive measures, and high rates of inappropriate VTE prophylaxis prescribing contribute to the gap between VTE prophylaxis and guidelines. To further minimize the gap between clinical practice and guidelines, a range of strategies have been employed across various fields of VTE prophylaxis. One of the most effective measures is the utilization of a Clinical Decision Support System (CDSS). Smart technology-based CDSS facilitates automated evaluation of VTE risk and detection, addressing issues at both the beginning and end of the in-hospital VTE prevention process. but there is still a lack of research on how to effectively implement evidence-based VTE prophylaxis in the middle of the process.

In our hospital, routine use of DeVTEcare system (a CDSS for VTE risk assessment and integrated care) for in-hospital management of VTE has been launched since 2021. This study aims to investigate the effect of integrating bundled guideline-based VTE prevention strategies into the DeVTEcare system on in-hospital VTE prophylaxis.

ELIGIBILITY:
Inclusion Criteria:

* Discharged patients who were ≥18 years of age at admission were included in the observation cohort. If a patient had multiple hospitalizations, information on only the longest hospitalization was included in the study.

Exclusion Criteria:

* Lack of diagnostic information；
* Length of hospitalization ≤ 24 hours；
* Patients on anticoagulation therapy at the time of admission: e.g., those with established VTE, atrial fibrillation, acute myocardial infarction, ischemic stroke, those on continuous renal replacement therapy, extracorporeal membrane pulmonary oxygenation, hemodialysis, and mechanical valve implantation status.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: In our hospital, routine use of DeVTEcare system (a CDSS for VTE risk assessment and integrated care) for in-hospital management of VTE has been launched since 2021. By retrospectively collecting information on discharged patients, all patients discharged from our hospital between April 2023 and April 2024 will be included in the pre-modified DeVTEcare group.
  The modified DeVTEcare system, which incorporates bundled guideline-based VTE prevention measures, will be utilized to assist healthcare providers in VTE prophylaxis after September 2024. By retrospectively collecting information on discharged patients, all patients discharged from our hospital between September 2024 and February 2025 will be included in the post-modified DeVTEcare group.
Sampling Method: Non-Probability Sample
Enrollment: 15626 (Estimated)
Dates: Start 2024-09-01 (Estimated); Primary Completion 2025-02-28 (Estimated); Study Completion 2025-02-28 (Estimated)

PRIMARY OUTCOMES:
In-hospital VTE | During the hospitalization (assessed up to 30 days)
  In-hospital VTE refers to the occurrence of a VTE in a patient who did not have a VTE on admission but developed one during the course of their hospital stay.

SECONDARY OUTCOMES:
Guideline-compliant prescription of VTE prophylaxis | During the hospitalization (assessed up to 30 days)
  Guideline-compliant prescription of VTE prophylaxis refers to the adoption of risk stratification to guide clinicians' decisions to prescribe guideline recommended thromboprophylaxis.
Preventable VTE | During the hospitalization (assessed up to 30 days)
  Preventable VTE is defined as occurring in a high-risk patient not prescribed adequate VTE prophylaxis.
Hospital-related VTE death | During the hospitalization (assessed up to 30 days)
  Hospital-related VTE death is defined as patient who died during the present hospitalization while having an in-hospital VTE event.
Major bleeding | During the hospitalization (assessed up to 30 days)
  The major bleeding events are defined by the International Society on Thrombosis and Hemostasis (ISTH) and are further categorized into VTE prophylaxis-related major bleeding and VTE treatment-related major bleeding.
Non-major bleeding | During the hospitalization (assessed up to 30 days)
  The non-major bleeding events are defined by the International Society on Thrombosis and Hemostasis (ISTH) and are further categorized into VTE prophylaxis-related non-major bleeding and VTE treatment-related non-major bleeding.

CONTACTS AND LOCATIONS:
Overall Officials: ZHI-GENG JIN, Doctor, Study Chair — Sixth Medical Center of Chinese PLA General Hospital

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Henke PK, Kahn SR, Pannucci CJ, Secemksy EA, Evans NS, Khorana AA, Creager MA, Pradhan AD; American Heart Association Advocacy Coordinating Committee. Call to Action to Prevent Venous Thromboembolism in Hospitalized Patients: A Policy Statement From the American Heart Association. Circulation. 2020 Jun 16;141(24):e914-e931. doi: 10.1161/CIR.0000000000000769. Epub 2020 May 7. PMID 32375490
- [Background] Jin ZG, Zhang H, Tai MH, Yang Y, Yao Y, Guo YT. Natural Language Processing in a Clinical Decision Support System for the Identification of Venous Thromboembolism: Algorithm Development and Validation. J Med Internet Res. 2023 Apr 24;25:e43153. doi: 10.2196/43153. PMID 37093636
- [Background] Durieux P, Nizard R, Ravaud P, Mounier N, Lepage E. A clinical decision support system for prevention of venous thromboembolism: effect on physician behavior. JAMA. 2000 Jun 7;283(21):2816-21. doi: 10.1001/jama.283.21.2816. PMID 10838650